CLINICAL TRIAL: NCT00567788
Title: Comparison of Bimatoprost and Lataprost in Patients With Chronic Angle-Closure Glaucoma: A Randomized Cross-Over Study
Brief Title: Comparison of Bimatoprost and Latanoprost in Patients With Chronic Angle-Closure Glaucoma: A Randomized Cross-Over Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Singapore National Eye Centre (Other Government)
Collaborators: Allergan (Industry)
Responsible Party: Aung Tin, Singapore National Eye Centre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R353/11/2004; SQGL08
Record Dates: First submitted 2007-12-04; First posted 2007-12-05 (Estimated); Last update posted 2007-12-05 (Estimated); Status verified 2007-11

CONDITIONS: Glaucoma, Angle-Closure
Keywords: Glaucoma, angle-closure
MeSH Terms: conditions — Glaucoma, Angle-Closure | interventions — Latanoprost; Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Study subjects will be randomized to receive either latanoprost once daily or bimatoprost once daily for 6 weeks, after which they will be crossed over to the other medication for another 6 weeks. The IOP-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Interventions: Drug: Latanoprost-Bimatoprost
- 2 (Active Comparator): Study subjects will be randomized to receive either latanoprost once daily or bimatoprost once daily for 6 weeks, after which they will be crossed over to the other medication for another 6 weeks. The IOP-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline.
  Interventions: Drug: Bimatoporost-Latanoprost

INTERVENTIONS:
Drug: Latanoprost-Bimatoprost — latanoprost 0.005% once daily followed by bimatoprost 0.03%
  Other Names: Xalatan, Lumigan
  Arms: 1
Drug: Bimatoporost-Latanoprost — bimatoprost 0.03% once daily followed by latanoprost 0.005%
  Other Names: Xalatan, Lumigan
  Arms: 2

SUMMARY:
This is a randomized observer-masked cross-over study to compare the intraocular pressure (IOP) reducing effect of latanoprost with bimatoprost in subjects with chronic angle closure glaucoma (CACG) with raised IOP. Study subjects will be randomized to receive either latanoprost once daily or bimatoprost once daily for 6 weeks, after which they will be crossed over to the other medication for another 6 weeks. The IOP-reducing effect of the medications will be assessed by the reduction in IOP after each medication compared to baseline. The study will be carried out in at least 2 Singapore hospitals.

DETAILED DESCRIPTION:
Study eyes are defined as the eye(s) that fulfil all inclusion criteria but none of the exclusion criteria. The IOP will be measured by Goldmann applanation tonometry. The IOP at every visit will be taken by one examiner (masked) using the same slit lamp and tonometer. Three consecutive readings will be taken at each time and the mean of the three values used in the statistical analysis. The examiner will not be aware of the treatment the patient is on. The scale of the tonometer will be concealed to the examiner, and the IOP value read off by an assistant after the examiner determines the end point of tonometry.

At the Baseline visit and last visit of each Treatment period (Day 0, 42 and 84), IOP will be measured at 9 am and 5 pm. On Day 14 and 56, IOP will be measured only at 9 AM.

Thus, when the IOP is measured in the clinic at 9 AM, approximately 13 hours would have elapsed from the evening dose. This will coincide with the approximate peak effect of bimatoprost and latanoprost. The IOP reading at 5 PM will be the approximate trough for latanoprost and bimatoprost.

The IOP at the end of each Treatment period at 6 weeks (Day 42 and 84) will be utilized as the primary endpoint and a comparison of mean IOPs of the two treatment groups compared with the baseline (Day 0). For those who do not, for any reason, complete the 6-week assessment, their last IOP measure will be carried forward to provide the endpoint. However, the number of such cases within each treatment group will also be reported.

Prior to the trial, all patients will undergo clinical examinations and eye tests to determine eligibility.

After being enrolled into the trial, patients will be randomized to receive either latanoprost or bimatoprost. They will be subjected to a list of tests (details of schedule and procedures in Appendix A) on the baseline day (Day 0) and instructed that the first eye application will start at 8pm on the same day. For 6 weeks, patients assigned to the latanoprost treatment group will administer latanoprost 0.005% in the evening. Patients assigned to the bimatoprost group will administer 0.03% bimatoprost once daily (in the evening). Study visits will be on Day 14 (Visit 2) and Day 42 (Visit 3).

After 6 weeks, patients will be crossed over to the other medication. Patients will undergo exactly the same regimen of examination and clinic visits as in Treatment period I. Study visits will be on Day 56 (Visit 4) and Day 84 (Visit 5).

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral or bilateral CACG
2. Age more than or equal to 40 years old
3. Informed consent obtained at pre-study visit for all patients

Exclusion Criteria:

1. Secondary glaucoma such as uveitic or neovascular glaucoma
2. One eye eligible and fellow eye on unsuitable glaucoma treatment for this trial
3. IOP > 36 mmHg at Pre-study visit
4. Advanced glaucoma at risk of progression. This is defined as vertical cup-disc ratio > 0.9 and/or central visual field loss with a sensitivity of < 10 dB in any of the 4 visual field test points closest to fixation
5. Ocular infection or inflammation (except when related to peripheral iridotomy) within 3 months of the prestudy visit
6. On more than two anti-glaucoma medications
7. Previous intraocular surgery apart from laser peripheral iridotomy
8. Previous trauma to the eye, with angle damage
9. Ocular treatment with a steroid or non-steroidal anti-inflammatory medication within 1 month of the prestudy visit.
10. Use of contact lens.
11. Cornea infection or other cornea abnormalities.
12. Ocular diseases such as dry eye or retinal pathology.
13. Oral medications, such as diuretics, known to affect IOP.
14. Cerebrovascular, hepatic, renal, metabolic disease.
15. Known allergy to benzalkonium, or any other components of latanoprost/bimatoprost.
16. History of non-compliance.
17. Women who are pregnant, lactating, or of childbearing potential and not using adequate contraception.
18. Participated in another therapeutic medication study within the last 1 month.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-07; Study Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint is defined as IOP reduction from baseline measurement (week 0) to the measurement at week 6 at each treatment period. | 6 weeks

SECONDARY OUTCOMES:
Incidence of side effects of each medication. | 6 weeks after each treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Tin Aung, Principal Investigator — SNEC
Locations (1):
- Singapore National Eye Centre, Singapore, Singapore